CLINICAL TRIAL: NCT02100033
Title: How Acupuncture Sensation Propagated to Effect the Energy of Channels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CMUH102-REC1-090
Record Dates: First submitted 2014-03-17; First posted 2014-03-31 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Acupuncture Manipulation
MeSH Terms: interventions — Acupuncture Therapy

ARMS (1):
- acupuncture (Experimental): acupuncture manipulation
  Interventions: Device: acupuncture

INTERVENTIONS:
Device: acupuncture

SUMMARY:
De-qi as an important factor to therapeutic effect of acupuncture for years, It's a concrete pathway to approach Qi, an abstract concept in Chinese medicine. However, all previous physicians and medical scientists have different interpretation to De-qi, and no objective principles for clinical practice, teaching and studies.

Qi propagated combined with acupuncture practice always be seen as De-qi , therefore, the study control "transmission or not" and "direction of sensation propagated" to compare what's different in human body. If the change happened as prediction based on acupuncture theories, it could define De-qi for operation.

The study will collect 60 subjects, from age 20 to 40, the same numbers of male and female. They will accept different manipulation in left hand HeGu(LI4), and assessed the variations in microcirculation, temperature of left forearm, and waxing/waning of yin-yang , Qi and blood in related meridian. We hope to understand if sensation propagated is primary factor of De-Qi and acupuncture effect .

ELIGIBILITY:
Inclusion Criteria:

* both male and female
* age:20-40 years old

Exclusion Criteria:

* to be afraid of acupuncture
* easily fainting
* right index finger has been injured recent one month
* had taken drugs can trigger vasodilatation or vasoconstriction recent three months
* systemic diseases
* pregnancy

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
variation trend of electric conductivity | 30-60seconds per trial

SECONDARY OUTCOMES:
blood flow speed | 30-60seconds per trial

OTHER OUTCOMES:
EEG | 30-60seconds per trial

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan